CLINICAL TRIAL: NCT04824157
Title: Ketamine IV Classic Protocol : Five Years Follow up Clinical Evaluation.
Brief Title: Ketamine IV Classic Protocol : Five Years Follow up
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Revital Amiaz, Head of Department Psychiatry B, Sheba Medical Center
Other Study IDs: 5826-18-SMC
Record Dates: First submitted 2019-12-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Major Depressive Disorder; Drug Abuse; Medications; Relapse
Keywords: Major depressive disorder; ketamine; follow up; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Substance-Related Disorders; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non — Follow up

SUMMARY:
Patients who suffer from MDD recieved ketamnie (2014-15) in open study will be addressed and there depression mood will be evaluated using the rating scale that were used in the original research. In addition time of relapse and questions about their medications and drug use will be performed.

DETAILED DESCRIPTION:
Patients who suffer from Major Depressive disorder and are outpatients in our clinic and, received in the years (2014-15) ketamine in open study will be addressed and there depression mood will be evaluated using the rating scale that were used in the original research. In addition time of relapse and questions about their medications and drug use will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient who participated in ketamine study 1126

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who participated in ketamine study 1126 and are willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Mood that will be evaluated using the MADRAS Montgomery-Asberg Depression Rating Scale". | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data with other resarchers that will be interested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to 6 weeks from demand
Access Criteria: Six weeks